CLINICAL TRIAL: NCT05055648
Title: PROton Versus Photon Therapy for Esophageal Cancer - a Trimodality Strategy (PROTECT) a Multicenter International Randomized Phase III Study of Neoadjuvant Proton Versus Photon Chemoradiotherapy in Locally Advanced Esophageal Cancer
Brief Title: PROton Versus Photon Therapy for Esophageal Cancer - a Trimodality Strategy
Acronym: PROTECT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Leeds (Other); KU Leuven (Other); University College, London (Other); Aarhus University Hospital (Other); Technische Universität Dresden (Other); Academisch Ziekenhuis Groningen (Other); CNAO National Center of Oncological Hadrontherapy (Other); Agenzia Nazionale per i Servizi Sanitari Regionali (Other); Centre Antoine Lacassagne (Other); Centre Leon Berard (Other); Institut Curie (Other); Maastro Clinic, The Netherlands (Other); University College London Hospitals (Other); The Christie NHS Foundation Trust (Other); Paul Scherrer Institut, Center for Proton Therapy (Other); HollandPTC (Industry); IBA worldwide (Unknown); Varian- A Siemens Healthineer Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCPT101008134
Record Dates: First submitted 2021-08-26; First posted 2021-09-24 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer; Radiotherapy; Side Effect; Proton Therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: open-label, non-blinded, international multicenter, randomized phase III study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photon Arm (Active Comparator): Standard arm with neoadjuvant chemoradiotherapy (nCXT) with photons
  Interventions: Radiation: Photon Radiotherapy
- Proton Arm (Experimental): Experimental arm with neoadjuvant chemoradiotherapy (nCPT) with protons
  Interventions: Radiation: Proton Radiotherapy

INTERVENTIONS:
Radiation: Photon Radiotherapy — nCXT consists of weekly carboplatin and paclitaxel for 5 weeks, following the CROSS trial. The radiation dose will be either 41.4 Gy in 23 fractions or 50.4 Gy in 28 fractions
  Arms: Photon Arm
Radiation: Proton Radiotherapy — nCPT consists of weekly carboplatin and paclitaxel for 5 weeks, following the CROSS trial. The radiation dose will be either 41.4 Gy in 23 fractions or 50.4 Gy in 28 fractions
  Other Names: Proton Therapy
  Arms: Proton Arm

SUMMARY:
The PROTECT trial will test the hypothesis that proton (PT) -enabled radiation dose reductions to sensitive, normal tissues will result in lower rates of treatment-related pulmonary complications in esophageal cancer compared to standard photon therapy (XT).

DETAILED DESCRIPTION:
PROTECT is a unblinded international multicenter randomized phase III study for patients with operable EC or EGC receiving nCXT (standard of care) or nCPT (intervention). The study will be open-label for the patient and the treating physician.

The radiation dose is either 41.4 Gy in 23 fractions, five fractions per week or 50.4 Gy in 28 fractions, five fractions per week. Prior to trial opening, each proton center will determine a single dose regimen for all patients treated in that specific proton center and its assigned photon centers.

The protocol prescribes that all referring centers will use the same chemotherapy regimen, which is weekly carboplatin (AUC 2), and paclitaxel (50 mg/m2), five cycles, irrespective of choice of dose regimen. Chemotherapy is a non-investigational drug.

Prior to referral to any proton therapy center, patients will be randomed (1:1) to either nCXT or nCPT. Only patients randomized to the PT arm will be referred to a PT center. Randomization will be performed centrally using an online 24-hour web-based system maintained by the Clinical Trial Office at Aarhus University Hospital, ensuring allocation concealment to the clinical investigators. The method of randomization will be stratified permuted blocks of size 4 and 6 (selected randomly) with the following strata:

* Histopathology (non-squamous vs squamous cell carcinoma)
* Planned surgical technique (open versus minimal invasive/robotic or hybrid)
* Proton center and sites assigned to this center (which will deliver the nCXT)

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified squamous cell carcinoma or adenocarcinoma (including signet cell carcinoma and large cell carcinoma, not further specified) of the esophagus (E) or gastro-esophageal junction (GEJ).

  * FDG PET/CT performed.
  * Tumor stage according to TNM (8th edition): cT1-4a and/or cN+, cM0.
  * Age ≥18 years.
  * Performance status WHO ≤2.
  * Adequate laboratory findings: hematological: hemoglobin > 90 g/L, absolute neutrophil count (ANC) ≥ 1,5 x 109/L, platelets ≥ 75 x 109/L hepatic: bilirubin ≤ 1.5 x upper limit of normal (ULN), ALAT ≤ 3 x ULN renal: creatinine ≤ 1.5 x ULN, GFR (may be calculated) > 30 ml/min
  * MDT decision on suitability to undergo curatively intended nCXT or nCPT followed by surgery.
  * Planned transthoracic esophagectomy or gastrectomy being open, minimally invasive of combination of both.
  * Ability to adhere to procedures for study and follow-up.
  * Patients with low risk cancers with a life expectancy above 5 years (e.g. low risk prostate cancer) are allowed in the study. Adequately treated diagnoses such as cervix uteri carcinoma in situ, in situ urothelial carcinoma or localized non-melanoma skin cancer are allowed, regardless of time of diagnosis.
  * Patients of childbearing potential: pregnancy prevention according to the standards of each country. Patients of childbearing potential must present a negative pregnancy test. Patients and their partners must use effective contraception. Patients of childbearing potential included in the study must use oral contraceptives, intrauterine devices, depot injection of progestin subdermal implantation, a hormonal vaginal ring, or transdermal patch during the study treatment and one month after.

Exclusion Criteria:

Patients who meet one or more of the following exclusion criteria cannot be included in the study:

* Prior thoracic XT or PT, chemotherapy or surgical resection in the esophageal/gastric region (previous EMR or ESD is allowed).
* Tumor < 3 cm from oropharyngeal sphincter.
* Planned transhiatal resection
* Patients with other previous malignancies are excluded unless a complete remission or complete resection was achieved at least 5 years prior to study entry.
* Any unstable systemic disease (including clinically significant lung and cardiovascular disease, unstable angina, New York Heart Association (NYHA) grade III-IV congestive heart, severe hepatic, renal or metabolic disease or active inflammatory bowel disease).
* Symptomatic peripheral neuropathy greater than grade 1 (scored according to CTCAE v5.0).
* Any other serious or uncontrolled illness, which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial.
* Unable to understand and digest study patient information or comply with study treatment and safety instructions.
* Gastro-esophageal stent within the irradiated volume.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary complications | from randomization until 90 days after surgery
  Incidence of pulmonary complications during and following nCPT or nCXT and surgery

SECONDARY OUTCOMES:
Early toxicity | from start of nCPT or nCXT until surgery
  Predefined items ≥ grade 2 scored by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Late toxicity | up to 5 years
  Predefined items ≥ grade 2 scored by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Postoperative complications | from surgery until 90 days after surgery
  Predefined items scored by Clavien-Dindo and Comprehensive Complications Index (CCI)
Major cardiovascular events (MACE) | up to 5 years
  Predefined cardiovascular events scored by MACE
Patient-reported outcome measures | up to 5 years
  EORTC quality of life questionnaire
Compliance with trimodality treatment | 3 months
  The proportion of patients complying with trimodality treatment in each arm
Pathological response | immediately after surgery
  tumor regression grade for the primary tumor scored according to Mandard score.
Cumulative incidence of loco-regional failure | from date of randomization up to 5 years
  Locoregional failure evaluated according to RECIST with all failures within the irradiated volume counting as events.
Pattern of failure | up to 5 years
  First site of failure will be divided in loco-regional lymph node failures, loco-regional failures in anastomosis, and distant extra-cranial and intra-cranial failures. All loco-regional failures will be divided in failures inside and outside the treatment volume, which is defined to be within the specified treatment dose.
Disease-free survival (DFS) | up to 5 years
  Disease control evaluated according to RECIST with any recurrence (locoregional or distant) as well as death from any cause, whatever occurs first, will be considered as events.
Overall survival (OS) | up to 5 years
  Death from all causes will considered as events

OTHER OUTCOMES:
Total toxicity burden (TTB) | from randomization until 90 days after surgery
  The combined toxicity scale TTB used in the trial by Lin et al (Lin 2020)
Concordance of observed pulmonary complications with predicted complications from NTCP models | up to 5 years
  Comparison of observed and predicted toxicity rates
Blood biomarkers as predictors for treatment failure | up to 5 years
  circulating tumor DNA
Proportion of patients receiving adjuvant immunotherapy | up to 5 years
  The actual number of patients starting adjuvant immunotherapy will be recorded
Cost-effectiveness of proton therapy relative to photon therapy | up to 5 years
  Incremental cost effectiveness ratios (ICERs), cost per QALY gained, cost per complication avoided, and cost per total toxicity burden avoided will be reported.
FDG/PET CT as predictors for treatment failure | 12 months
  Correlation between diagnostic PET, planning PET-CT and PET at 12 months
Concordance of observed cardiac complications with predicted | Up to 5 years
  Comparison of observed and predicted toxicity rates

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Nordsmark, Dr., Study Director — University of Aarhus; Karin Haustermans, Dr., Study Chair — UKleuven
Locations (15):
- Catholic University of Leuven, Leuven, Belgium
- Aarhus University Hospital (AUH), Aarhus, Denmark
- France (3):
  - Centre Léon Bérard (CLB), Lyon
  - Centre Antoine Lacassagne (CAL), Nice
  - Institut Curie, Paris
- Technische Universität Dresden (TUD), Dresden, Germany
- Italy (3):
  - San Raffaele Hospital, Milan
  - Centro Nazionale di Adroterapia Oncologica (CNAO), Pavia
  - Azienda Provinciale Per I Servizi Sanitari (APSS), Trento
- Netherlands (2):
  - Academisch Ziekenhuis Groningen (UMCG), Groningen
  - Stichting Maastricht Radiation Oncology (MAASTRO), Maastricht
- Switzerland (2):
  - Paul Scherrer Institute (PSI), Villigen
  - University Hospital Zurich (USZ), Zurich
- United Kingdom (2):
  - University College London Hospital (UCLH), London
  - The Christie NHS foundation trust, Manchester

IPD SHARING:
Plan to Share IPD: No